CLINICAL TRIAL: NCT00089284
Title: A Phase I/II Trial of Redox Regulation in Patients With Relapsed or Refractory CD20 Positive Non-Hodgkin's Lymphoma (NHL): Combining 90-Yttrium- Zevalin and the Redox- Modulating Agent, Motexafin Gadolinium (MGd)
Brief Title: Phase I/II Trial of Redox Regulation in Patients With Relapsed or Refractory CD20+ NHL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to lack of funding, phase II of study was not completed.
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 02H8; 1346001 (Other: Northwestern University IRB)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-04

CONDITIONS: Non-Hodgkin's Lymphoma (NHL)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; motexafin gadolinium; Injections; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituxan and 90Yttrium-Zevalin plus MGd (Experimental): Patients receive motexafin gadolinium IV over 30-60 minutes on days 1-4 and 8-11. At least 1 hour after motexafin gadolinium administration, patients receive rituximab IV over 3-4 hours on days 1 and 8. After rituximab administration, patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1. Patients undergo gamma camera scanning on days 1, 2*, 4*, and 7 and dosimetry on days 2, 4, and 7. If safe biodistribution is demonstrated, patients receive yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes (after rituximab administration) on day 8.
  Interventions: Drug: Rituxan; Drug: motexafin gadolinium; Drug: 111Indium-Zevalin and 90Yttrium-Zevalin

INTERVENTIONS:
Drug: Rituxan — Patients receive motexafin gadolinium IV over 30-60 minutes on days 1-4 and 8-11. At least 1 hour after motexafin gadolinium administration, patients receive rituximab IV over 3-4 hours on days 1 and 8. After rituximab administration, patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1. Patients undergo gamma camera scanning on days 1, 2*, 4*, and 7 and dosimetry on days 2, 4, and 7. If safe biodistribution is demonstrated, patients receive yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes (after rituximab administration) on day 8.
  Other Names: rituximab IDEC-C2B8
Drug: motexafin gadolinium — Patients receive motexafin gadolinium IV over 30-60 minutes on days 1-4 and 8-11. At least 1 hour after motexafin gadolinium administration, patients receive rituximab IV over 3-4 hours on days 1 and 8. After rituximab administration, patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1. Patients undergo gamma camera scanning on days 1, 2*, 4*, and 7 and dosimetry on days 2, 4, and 7. If safe biodistribution is demonstrated, patients receive yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes (after rituximab administration) on day 8.
  Other Names: MGd, Xcytrin® (motexafin gadolinium) Injection,; NSC 695238
Drug: 111Indium-Zevalin and 90Yttrium-Zevalin — Patients receive motexafin gadolinium IV over 30-60 minutes on days 1-4 and 8-11. At least 1 hour after motexafin gadolinium administration, patients receive rituximab IV over 3-4 hours on days 1 and 8. After rituximab administration, patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1. Patients undergo gamma camera scanning on days 1, 2*, 4*, and 7 and dosimetry on days 2, 4, and 7. If safe biodistribution is demonstrated, patients receive yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes (after rituximab administration) on day 8.
  Other Names: Ibritumomab-tiuxetan

SUMMARY:
Monoclonal antibodies such as rituximab and yttrium Y 90 ibritumomab tiuxetan can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells. Motexafin gadolinium may increase the effectiveness of yttrium Y 90 ibritumomab tiuxetan by making the cancer cells more sensitive to the drug.

This phase I/II trial is studying the side effects and best dose of motexafin gadolinium when administered with rituximab and yttrium Y 90 ibritumomab tiuxetan and to see how well they work in treating patients with stage II, stage III, or stage IV relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
This is a phase I, dose-escalation study of motexafin gadolinium followed by a phase II study. Patients are stratified according to extent of lymphomatous involvement (≤ 5% vs > 5 but ≤ 24% of cellular elements).

Cohorts of 3-6 patients in each stratum receive escalating doses of motexafin gadolinium until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity (DLT) OR the dose preceding that at which 2 of 3 or 3 of 6 patients experience DLT.

* Once the MTD is determined, additional patients are treated at that dose level as in phase I.

Patients are followed weekly for 3 months and then monthly for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one of the following:

  * Low-grade or follicular B-cell non-Hodgkin's lymphoma (NHL)

    * The following histologies are eligible:

      * Small lymphocytic lymphoma
      * Lymphoplasmacytoid lymphoma
      * Follicular center grades 1, 2, or 3 lymphoma
      * Extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue type
      * Nodal marginal zone B-cell lymphoma
    * Relapsed or refractory after 2 prior treatment regimens or 1 anthracycline regimen
  * Diffuse large B-cell NHL or mantle cell lymphoma in first or second relapse
  * Transformed NHL, defined as low-grade NHL transformed to diffuse large B-cell lymphoma, with no more than 1 relapse since transformation

Age 18 and over Recovered from prior immunotherapy Life expectancy At least 3 months Recovered from prior chemotherapy

* More than 4 weeks since prior major surgery and recovered
* More than 4 weeks since prior anticancer therapy recovered from prior radiotherapy

Exclusion criteria:

No major bleeding within the past 4 weeks No uncontrolled hypertension No stroke within the past 4 weeks

* No active infection
* No other active nonmalignant disease
* No known G6PD deficiency
* No history of porphyria
* No other condition that would preclude study participation
* No human anti-mouse antibodies
* No known history of HIV
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior radioimmunoconjugate therapy
* No prior exposure to murine antibodies other than rituximab
* More than 4 weeks since prior rituximab
* No history of failed stem cell collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-10-28 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2008-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M. Evens, DO, MS, Principal Investigator — Northwestern University; Leo I. Gordon, MD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Jesse B. Brown Veterans Affairs Medical Center, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to accrual between the dates of September 10, 2003 and October 31, 2007 with the first patient enrolled on study October 28, 2003. Patients were recruited from the outpatient Hematology-Oncology clinic at Northwestern Medical Faculty Foundation, and the in-patient Hematology-Oncology service of Northwestern Memorial Hospital.
Pre-assignment Details: For phase I, patients were allocated according to the amount of bone marrow involvement they expressed (either ≤ 5% or ≤ 6-24% involvement). Initially, patients were accrued to the first cohort of the ≤ 5% involvement group. After that group moved to the second cohort, patients in the ≤ 6-24% involvement group were enrolled to the first cohort.
Groups:
- Phase I: 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement: For the phase I dose-escalation portion, patients were allocated based on the amount of lymphoma bone marrow involvement. Initially, enrollment to the first cohort (2.5 mg/kg MGd) was open only to those with ≤ 5% of bone marrow involvement.
- Phase I: 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement: In the phase I portion of the study, following completion of enrollment of patients with ≤ 5% bone marrow involvement to their first cohort (2.5 mg/kg MGd), patients with 6-24% bone marrow involvement could be enrolled to their first cohort (2.5 mg/kg MGd).
- Phase I: 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement: After completion of the first cohort (2.5 mg/kg MGd) in the ≤ 5% Bone Marrow Involvement group, patients with ≤ 5% Bone Marrow Involvement were enrolled to the second cohort (3.5 mg/kg MGd).
- Phase I: 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement: After completion of the second cohort (3.5 mg/kg MGd) in the ≤ 5% Bone Marrow Involvement group, patients with ≤ 5% Bone Marrow Involvement were enrolled to the third cohort (5.0 mg/kg MGd).
- Phase I: 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement: After completion of the first cohort (2.5 mg/kg MGd) in the ≤ 6-24% Bone Marrow Involvement group, patients with ≤ 6-24% Bone Marrow Involvement were enrolled to the second cohort (3.5 mg/kg MGd).
- Phase I: 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement: After completion of the second cohort (3.5 mg/kg MGd) in the ≤ 6-24% Bone Marrow Involvement group, patients with ≤ 6-24% Bone Marrow Involvement were enrolled to the third cohort (5.0 mg/kg MGd).
- Phase II: 5.0 mg/kg MGd & </= 5% Bone Marrow Involvement: After completion of the Phase I portion, patients were enrolled to the maximum tolerated dose (MTD) group of 5.0 mg/kg MGd for </+ 5% Bone Marrow Involvement.
Period: Overall Study
Arm/Group | Phase I: 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase I: 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase I: 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase II: 5.0 mg/kg MGd & </= 5% Bone Marrow Involvement
Started | 7 | 3 | 6 | 6 | 0 (No patients were accrued to this cohort of 6-24% involvement due to lack of eligible patients.) | 0 (No patients were accrued to this cohort of 6-24% involvement due to lack of eligible patients.) | 8
Completed | 7 | 3 | 6 | 6 | 0 | 0 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse event before starting treatment | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase I: 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase II: 5.0 mg/kg MGd & </= 5% Bone Marrow Involvement | Total
Number analyzed (Participants) | 7 | 3 | 6 | 6 | 8 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 3 | 4 | 4 | 17
  >=65 years | 3 | 1 | 3 | 2 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 2 | 5 | 15
  Male | 4 | 1 | 3 | 4 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants] — All patients were assigned race at the time of registration according to how their race is listed in their medical records.
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
    Asian | 0 | 0 | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    White | 6 | 3 | 5 | 6 | 8 | 28
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 6 | 6 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities (DLT)
Description: The number of Dose Limiting Toxicities (DLT) observed in patients treated with Motexafin Gadolinium at different dose levels in combination with Rituxan, Indium-Zevalin, and 90Yttrium-Zevalin was used to determine the Maximum Tolerated Dose (MTD) to be used for phase II of the study. The number of dose-limiting toxicities observed in each cohort of patients determined whether to continue dose escalation. Each cohort = at least 3 patients.
  All toxicities will be graded according to the NCI Common Toxicity Criteria, version 2.0, with a DLT defined as any of the following:
  Grade 3 or 4 non-hematologic toxicity (other than grade 3 nausea or vomiting). Grade 4 vomiting despite maximal antiemetic support. Grade 4 neutropenia and thrombocytopenia either lasting longer than 14 days-Grade 4 duration will be measured (in days) from the first date in grade 4 to last date in grade 4 after nadir (growth factor and transfusion independent, respectively).
Time Frame: Weekly during treatment and continuing up through Day 90
Population: Only patients enrolled during the phase I portion of this trial were analyzed for this outcome measure.
Measure: Number; unit: Dose-Limiting Toxicities
Groups:
- 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement: For the phase I dose-escalation portion, patients were allocated based on the amount of lymphoma bone marrow involvement. Initially, enrollment to the first cohort was open only to those with ≤ 5% of bone marrow involvement.
- 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement: In the phase I portion of the study, following completion of enrollment of patients with ≤ 5% bone marrow involvement to the first cohort on the Lesser Bone Marrow Involvement arm, patients with 6-24% bone marrow involvement could be enrolled to the first cohort in the Greater Bone Marrow Involvement arm.
- 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement: Following completion of enrollment to the first cohort, patients with ≤ 5% bone marrow involvement were then enrolled to the second cohort (3.5 mg/kg MGd).
- 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement: Following completion of enrollment to the second cohort, patients with ≤ 5% bone marrow involvement were then enrolled to the third cohort (5.0 mg/kg MGd).
- 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement: Following completion of enrollment to their first cohort, patients with 6-24% bone marrow involvement were then enrolled to their second cohort (3.5 mg/kg MGd).
- 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement: Following completion of enrollment to their second cohort, patients with 6-24% bone marrow involvement were then enrolled to their third cohort (5.0 mg/kg MGd).
Arm/Group | 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement | 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement | 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement | 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement
Number analyzed (Participants) | 7 | 3 | 6 | 6 | 0 | 0
Dose-Limiting Toxicities | 0 | 0 | 0 | 0 |  |

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose (MTD) of Motexafin Gadolinium in combination with Rituxan, Indium-Zevalin, and 90Yttrium-Zevalin was determined using a modified Fibonacci phase I study design (with patient allocation based on amount of lymphoma bone marrow involvement) and will be used in phase II of the study. The MTD will be that dose at which 0/3 or 1/6 patients or 2/9 experience a Dose Limiting Toxicity (DLT), with the next higher dose level provoking DLT in 2/3 or 3/6 or 4/9 patients.
Time Frame: Weekly during treatment and continuing up through Day 90
Population: Phase I arms were evaluable for this outcome measure.
Measure: Number; unit: mg/kg
Arm/Group | Rituxan and 90Yttrium-Zevalin Plus MGd
Number analyzed (Participants) | 22
mg/kg | 5.0

3. Secondary Outcome: Anti-lymphoma Efficacy
Description: To assess the anti-lymphoma efficacy of the combination of MGd and 90Yttrium-Zevalin therapy. Disease response to treatment was categorized as complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or complete response/unconfirmed (CRu). The overall response rate (ORR) was then calculated. The time to treatment failure (TTF), overall survival (OS), and duration of response were determined.
Time Frame: At 1, 3 and 6 months
Population: All phase I and phase II patients were evaluated for response to treatment (anti-lymphoma efficacy). For the cohort with ≤ 5% bone marrow involvement treated at the 5.0 mg/kg MGd dose, results are based on 6 phase I patients and 8 phase II patients. 2 patients were determined not to be evaluable as they did not reach response time points.
Measure: Count of Participants; unit: Participants
Arm/Group | 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement | 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement | 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement | 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement
Number analyzed (Participants) | 7 | 3 | 5 | 13 | 0 | 0
Participants
  Complete Response (CR) | 6 | 0 | 2 | 3 |  |
  Partial Response (PR) | 0 | 1 | 1 | 1 |  |
  Stable Disease (SD) | 0 | 1 | 2 | 5 |  |
  Progressive Disease (PD) | 1 | 0 | 0 | 3 |  |
  Complete Response/Uncofirmed (CRu) | 0 | 1 | 0 | 1 |  |

4. Secondary Outcome: Study and Describe the Bio-locationization of Motexafin Gadolinium (MGd) in Tumors Using MRIs
Description: To study the tumor-specific bio-localization of MGd in lymphoma through magnetic resonance imaging (MRI) in a subset of patients. The first 2 patients of each cohort will have MRI imaging to measure if signal intensity, a correlate for MGd uptake, is increased in known areas of lymphomatous involvement.
Time Frame: At baseline (pre-treatment) and on Day 4 of treatment
Population: Data was not collected for analysis of this outcome measure due to lack of funding.
Arm/Group | Phase I: 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase I: 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase I: 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase II: 5.0 mg/kg MGd & </= 5% Bone Marrow Involvement
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Correlative Laboratory Studies
Description: To explore correlative laboratory studies of MGd (ie, uptake of MGd by peripheral mononuclear cells, effect of MGd upon peripheral lymphocyte subset populations).
Time Frame: On Day 1 and 4
Population: Data not collected for analysis of this outcome measure.
Arm/Group | Phase I: 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase I: 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement | Phase I: 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase I: 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement | Phase II: 5.0 mg/kg MGd & </= 5% Bone Marrow Involvement
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected daily during the treatment period (Days 1 through 11), then weekly up to 30 days after the last dose of study treatment, and then monthly up to 90 days after the last dose of study treatment.
Description: 1 patient was withdrawn from the study without receiving any Zevalin (Y90) and thus was not considered evaluable for toxicity/adverse events.
Groups:
- 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement: For the phase I dose-escalation portion, patients were allocated based on the amount of lymphoma bone marrow involvement. Initially, enrollment to the first cohort (2.5 mg/kg MGd) was open only to those with ≤ 5% of bone marrow involvement.
- 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement: In the phase I portion of the study, following completion of enrollment of patients with ≤ 5% bone marrow involvement to their first cohort (2.5 mg/kg MGd), patients with 6-24% bone marrow involvement could be enrolled to their first cohort (2.5 mg/kg MGd).
- 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement: After completion of the first cohort (2.5 mg/kg MGd) in the ≤ 5% Bone Marrow Involvement group, patients with ≤ 5% Bone Marrow Involvement were enrolled to the second cohort (3.5 mg/kg MGd).
- 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement: After completion of the second cohort (3.5 mg/kg MGd) in the ≤ 5% Bone Marrow Involvement group, patients with ≤ 5% Bone Marrow Involvement were enrolled to the third cohort (5.0 mg/kg MGd).
- 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement: After completion of the first cohort (2.5 mg/kg MGd) in the ≤ 6-24% Bone Marrow Involvement group, patients with ≤ 6-24% Bone Marrow Involvement were enrolled to the second cohort (3.5 mg/kg MGd).
- 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement: After completion of the second cohort (3.5 mg/kg MGd) in the ≤ 6-24% Bone Marrow Involvement group, patients with ≤ 6-24% Bone Marrow Involvement were enrolled to the third cohort (5.0 mg/kg MGd).
Arm/Group | 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement | 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement | 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement | 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement | 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/3 | 2/6 | 4/13 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3 | 6/6 | 13/13 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement (N=7) | 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement (N=3) | 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement (N=6) | 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement (N=13) | 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement (N=0) | 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement (N=0)
Death - not otherwise specified (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Patient became deceased - no other information available.
Death due to disease progression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Patient experienced disease progression ultimately resulting in death.
Febrile neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection with grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction, GU: left ureter (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Patient had undergone stent replacement prior to registration on-study - event was determined to be related to that and not to study treatment.
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be unrelated to study - occurred when patient discontinuing heart medication which resulted in heart failure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 2.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement (N=7) | 2.5 mg/kg MGd & 6-24% Bone Marrow Involvement (N=3) | 3.5 mg/kg MGd & ≤ 5% Bone Marrow Involvement (N=6) | 5.0 mg/kg MGd & ≤ 5% Bone Marrow Involvement (N=13) | 3.5 mg/kg MGd & 6-24% Bone Marrow Involvement (N=0) | 5.0 mg/kg MGd & 6-24% Bone Marrow Involvement (N=0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 2 (2) | 4 (4) | 12 (12) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2 (2) | 0/0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Bilirubin (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (2) | 6 (6) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Creatinine (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Cytokine release syndrome (infusion reaction) (Investigations) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Attributed as related to study treatment.
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermal change: skin discoloration (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 5 (5) | 11 (11) | 0 (0) | 0 (0) — Skin turned a green color. Attributed as related to study treatment.
Dermatology - Other: blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
FEV1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2) | 5 (5) | 10 (10) | 0 (0) | 0 (0) — Attributed as probably related to study treatment.
Fever (in absence of infection) (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GGT (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hemorrhage - gums (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 6 (6) | 11 (11) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 3 (3) | 6 (6) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Infection (Infections and infestations) | 4 (4) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Insomnia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Leukocytes (Blood and lymphatic system disorders) | 7 (7) | 3 (3) | 5 (5) | 13 (13) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 6 (6) | 3 (3) | 5 (5) | 12 (12) | 0 (0) | 0 (0)
Mood alteration - anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 7 (7) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Neutrophils (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 4 (4) | 11 (11) | 0 (0) | 0 (0)
Pain - chest/thorax not otherwise specified (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain - dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain - headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Pain - lacrimal (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain - myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Pain - pelvic (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 7 (7) | 3 (3) | 5 (5) | 13 (13) | 0 (0) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Attributed as related to study treatment.
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal - Other (hematuria) (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sweating (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste alteration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Transaminases - AST/ALT (Hepatobiliary disorders) | 5 (5) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary rentention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) — Attributed as possibly related to study treatment.
Weight gain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight loss (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to a lack of adequate funding, we were unable to complete 2 of the secondary objectives for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes